CLINICAL TRIAL: NCT04647903
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-, Active-Controlled, 4 Period, 4 Way Crossover Study to Evaluate the Abuse Potential of Manipulated Abuse-Deterrent Dextroamphetamine Sulfate Immediate Release (ADAIR) Formulation Compared to Dextroamphetamine Sulfate Immediate Release When Administered Intranasally to Nondependent, Recreational Stimulant Users
Brief Title: Study to Evaluate the Abuse Liability, Pharmacokinetics, Safety and Tolerability of an Abuse-Deterrent d-Amphetamine Sulfate Immediate Release Formulation (ADAIR)
Acronym: SEAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vallon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAL-104
Record Dates: First submitted 2020-11-13; First posted 2020-12-01 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: ADHD; Narcolepsy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Narcolepsy | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Oral Placebo + Intranasal manipulated ADAIR (Experimental): Oral Placebo + Intranasal manipulated ADAIR 30 mg
  Interventions: Drug: ADAIR 10 mg IR tablets; Drug: Placebo
- Oral Placebo + Intranasal crushed dextroamphetamine sulfate (Active Comparator): Oral Placebo + Intranasal crushed dextroamphetamine sulfate IR 30 mg
  Interventions: Drug: d-amphetamine sulfate; Drug: Placebo
- Oral ADAIR + Intranasal Placebo (Experimental): Oral ADAIR 30 mg + Intranasal Placebo
  Interventions: Drug: Placebo
- Oral Placebo + Intranasal Placebo (Placebo Comparator): Oral Placebo + Intranasal Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADAIR 10 mg IR tablets — manipulated ADAIR 3x10mg
  Other Names: ADAIR
  Arms: Oral Placebo + Intranasal manipulated ADAIR
Drug: d-amphetamine sulfate — crushed d-amphetamine sulfate 3x10mg
  Other Names: dextroamphetamine sulfate
  Arms: Oral Placebo + Intranasal crushed dextroamphetamine sulfate
Drug: Placebo — placebo for oral and intranasal administration

SUMMARY:
This is a randomized, double-blind, double-dummy, placebo- and active-controlled 4 period, 4 way crossover study to assess the intranasal abuse potential of manipulated ADAIR formulation in nondependent, recreational stimulant users. The study will consist of an outpatient Screening Visit, an in clinic Qualification Phase, an in-clinic Treatment Phase, and an outpatient Follow-Up visit.

DETAILED DESCRIPTION:
VAL-104 is a phase 1, randomized, double-blind, double-dummy, placebo- and active-controlled 4 period, 4 way crossover study to assess the intranasal abuse potential of manipulated ADAIR formulation in nondependent, recreational stimulant users. The study objectives include assessing the pharmacodynamics (PD), pharmacokinetics (PK), safety and tolerability of manipulated ADAIR 30mg when compared to crushed d-amphetamine sulfate and placebo. The primary PD endpoint is mean maximum drug liking (Emax) on a bipolar 100mm visual analog scale.

A total of 64 subjects demonstrating a confirmed positive response to stimulants will enter the treatment phase. Safety will be assess via adverse events, vital signs, ECGs, clinical laboratory tests and Columbia Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers, 18 to 55 years of age inclusive
* Recreational drug abuse experience (>/= 10 times lifetime abuse of a CNS stimulant, >/= 1 abuse of CNS stimulant in the previous 3 months)
* Prior intranasal recreational drug abuse experience
* Body mass index (BMI) 18 to 33 kg/m2 inclusive

Exclusion Criteria:

* History of any significant disease or disorder
* History or current diagnosis of substance dependence (excluding caffeine and nicotine)
* Any confirmed significant allergic reactions against any drug, or multiple allergies in the judgement of the investigator
* Positive for hepatitis B, hepatitis C or HIV infection
* Pregnant or lactating women
* Participation in an investigational drug or device study within the last 30 days prior to Day 1 of the study
* Confirmed positive drug screening
* Positive alcohol breath test at screening / any Day -1
* Heavy smoker (> 20 cigarettes, > 8 pipefuls or > 8 cigars per day)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Drug Liking Emax Visual Analog Scale (VAS) | Up to 24 hours post-dose
  Peak effect for drug liking based on bipolar VAS from 0-100 scale

SECONDARY OUTCOMES:
Take Drug Again Emax VAS | Up to 24 hours post dose
  Peak effect for take drug again based on bipolar VAS from 0-100 scale
Overall Drug Liking Emax VAS | Up to 24 hours post dose
  Peak effect for overall drug liking based on bipolar VAS from 0-100 scale
Plasma concentrations (PK parameters) | Up to 36 hours post dose
  plasma concentrations of ADAIR and dextroamphetamine sulfate
Safety (adverse events) | Day 1 to Day 18
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whitaker, M, Study Director — Vallon Pharmaceuticals, Inc.
Locations (1):
- Vallon Investigational Site, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no IPD plan